CLINICAL TRIAL: NCT07106567
Title: The Effect Of Mediterranean Diet Education On Blood Pressure Levels And Quality Of Life Of Hypertensive Patiens
Brief Title: Mediterranean Diet And Blood Pressure In Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Hicran Yıldız, Prof.Dr., Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UludağU1
Record Dates: First submitted 2025-07-13; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Mediterranean Diet; Quality of Life
Keywords: Mediterranean diet; hypertension; quality of life; nutrition education; chronic disease management.; blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Quasi-experimental
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet education (Experimental): Mediterranean diet education
  Interventions: Behavioral: Mediterranean diet education
- Kontrol (Other)
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Mediterranean diet education — The General Information Form, Physical Activity Questionnaire, Perceived Stress Scale, SF-36 Quality of Life Scale, and Mediterranean Diet Adherence Scale will be administered to hypertensive patients at each interview (at 0, 1, and 3 months). The intervention group will be trained on the Mediterranean Diet at the first meeting.
  Arms: Diet education
Other: Control — The General Information Form, Physical Activity Questionnaire, Perceived Stress Scale, SF-36 Quality of Life Scale, and Mediterranean Diet Adherence Scale will be administered to hypertensive patients at each interview (at 0, 1, and 3 months).
  Arms: Kontrol

SUMMARY:
An experimental randomized controlled trial was conducted to evaluate the effects of Mediterranean diet education on blood pressure levels and quality of life in hypertensive patients. The sample size was determined using power analysis (n=70). Data were collected using a General Information Form, Physical Activity Questionnaire, Perceived Stress Scale, SF-36 Quality of Life Scale, and Mediterranean Diet Adherence Scale. Both groups were administered the questionnaire and blood pressure measurements at 0, 1, and 3 months. The first application was administered to the intervention group before the education session.

DETAILED DESCRIPTION:
The experimental randomized controlled trial was conducted to evaluate the effect of Mediterranean diet education on blood pressure levels and quality of life in hypertensive patients. The sample size was determined using power analysis (n=70). Patients who met the inclusion criteria were assigned to the experimental (n=35) and control (n=35) groups using a simple randomization technique. Data were collected using the General Information Form, Physical Activity Questionnaire, Perceived Stress Scale, SF-36 Quality of Life Scale, and Mediterranean Diet Adherence Scale. Surveys and blood pressure measurements were administered to both groups at 0, 1, and 3 months. The initial application for the intervention group was conducted before the education session. In data evaluation, percentages, means, independent t-tests, Pearson chi-square tests, Yates chi-square tests, repeated measures variance analysis (ANOVA), Pearson correlation tests, and Bonferroni tests were used.

ELIGIBILITY:
Inclusion Criteria:

* - Being between 18 and 60 years of age
* Being willing and able to participate in the study
* Being diagnosed with primary hypertension at least 6 months ago
* Being in the inactive group according to the International Physical Activity Questionnaire
* Having a score of 35 or below on the Perceived Stress Scale
* Being literate.

Exclusion Criteria:

* - Having changed their eating habits in the last year
* If the patient is a woman, they are pregnant
* Having been diagnosed with an eating disorder
* Having been diagnosed with a psychiatric diagnosis and/or receiving psychological support
* Being on antidepressants and/or steroids
* Being on any diet/receiving dietitian support
* Having been diagnosed with heart failure, chronic kidney disease (CHF), cirrhosis, gastrointestinal system (GIS), or endocrine disease
* Having been diagnosed with depression
* Being on enteral or parenteral nutrition
* Being a smoker
* Having a mental or communication disability that would prevent the patient from answering questions
* Having a body mass index of 30 or higher.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Mediterranean diet adherence level | 0th month (1st day), 1st month and 3rd month
  Mediterranean Diet Adherence Scale:The scale consists of 14 questions. Each question is scored 1 or 0, depending on the amount consumed, to calculate a total score. Total scores are used to determine dietary compliance: a score of ≤5 indicates low compliance, 6-9 indicates moderate compliance, and ≥10 indicates high compliance.
Quality of Life level | 0th month (1st day), 1st month and 3rd month
  SF-36 Quality of Life Scale: The scale consists of 36 questions and eight subscales. Each subscale is scored separately from 0 to 100. Higher scores indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Yıldız, Prof.Dr., Principal Investigator — Bursa Uludag Unversity
Locations (1):
- Dumlupınar Family Health Center, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individuals included in the study were informed that the data obtained would be used and published only within the scope of this study, on condition that their identities remained confidential.